CLINICAL TRIAL: NCT03432065
Title: A Pilot Study of Buspirone for the Treatment of Anxiety in Youth with Autism Spectrum Disorders
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was withdrawn due to competing research interests and slow recruitment.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Tolga A Ceranoglu, Medical doctor, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-P-002731
Record Dates: First submitted 2018-02-06; First posted 2018-02-13 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Autism Spectrum Disorder; Anxiety
Keywords: Autism Spectrum Disorders; Anxiety; Pervasive Developmental Disorders; Buspar; Buspirone
MeSH Terms: conditions — Autism Spectrum Disorder; Anxiety Disorders; Child Development Disorders, Pervasive | interventions — Buspirone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Buspirone (Experimental): Buspirone tablets will be administered twice daily, and will be titrated to a maximum daily dose of 60mg for 8 weeks.
  Interventions: Drug: Buspirone

INTERVENTIONS:
Drug: Buspirone — Children with autism spectrum disorders will receive buspirone treatment for eight weeks. Buspirone will be titrated to the maximum daily dose during the first four weeks of the trial (dose titration phase). Week 4 onwards, subjects will be maintained on maximum achieved dose until the end of the trial. During the titration phase, total dose will be increased by 10mg at each visit and by 5mg on the 4th day after each visit.

SUMMARY:
The main objective of this exploratory 8-week pilot study is to evaluate the safety and efficacy of buspirone for the treatment of anxiety in youth (ages 6-17 years) with autism spectrum disorders. The study results will be used to generate hypotheses for a larger randomized-controlled trial with explicit hypotheses and sufficient statistical power.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants between 6 and 17 years of age
* DSM-5 ASD diagnostic criteria as established by clinical diagnostic interview
* Participants with a score of ≥60 or more on the Anxiety/Depression subscale of CBCL
* Subjects can be taking psychotropic medications if they have been on the medication for at least 4 weeks prior to initiating study treatment and if they are on a stable dose, provided the medication is not listed in the Concomitant Medications section of the protocol.

Exclusion Criteria:

* History of active seizure disorder (EEG suggestive of seizure activity and/or history of seizure in last 1 month)
* Subjects with a medical condition or treatment that will either jeopardize subject safety or affect the scientific merit of the study, including:
* Pregnant or nursing females
* Organic brain disorders
* Uncorrected hypothyroidism or hyperthyroidism
* Clinically significant abnormalities on ECG (e.g., QT prolongation, arrhythmia)
* History of renal or hepatic impairment.
* Clinically unstable psychiatric conditions or judged to be at serious suicidal risk
* Current diagnosis of schizophrenia or bipolar disorder
* History of substance use (except nicotine or caffeine) within past 3 months or urine drug screen positive for substances of abuse
* Current treatment with medication with primary central nervous system activity (as specified in the Concomitant Medication section of the protocol)
* A non-responder or history of intolerance to buspirone, after treatment at an adequate dose and duration as determined by the clinician
* Subjects currently taking monoamine oxidase inhibitors (MAOI) and/or CYP3A4 inducers or inhibitors including nefazodone, diltiazem, verapamil, erythromaycin, itraconazole, or rifampin.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Reduction in Child and Adolescent Symptom Inventory-5-Anxiety (CASI-Anx) Score | Baseline to 8 Weeks
  The primary outcome measure of efficacy will be assessed by the reduction in anxiety symptom severity as measured by a change from baseline on the Child and Adolescent Symptom Inventory-5-Anxiety (CASI-Anx) scores. Responders are defined as those who demonstrate a >30% reduction on the CASI-Anx.

CONTACTS AND LOCATIONS:
Overall Officials: Atilla Ceranoglu, MD, Principal Investigator — Massachusetts General Hospital